CLINICAL TRIAL: NCT03715998
Title: A Phase 2, Double-blind, Active-controlled, Dose-titrating Efficacy and Safety Study of Firibastat Compared to Ramipril Administered Orally, Twice Daily, Over 12 Weeks to Prevent Left Ventricular Dysfunction After Acute MI
Brief Title: Firibastat or Ramipril After Acute Myocardial Infarction for Prevention of Left Ventricular Dysfunction
Acronym: QUORUM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Quantum Genomics SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QGC001-2QG4
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Results first posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2020-12

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Ramipril; firibastat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: firibastat 100 mg (Experimental): Subjects will receive 50 mg firibastat BID for 2 weeks and then 100 mg BID for 10 weeks.
  Interventions: Drug: Firibastat
- Group 2: firibastat 500 mg (Experimental): Subjects will receive 250 mg firibastat BID for 2 weeks and then 500 mg BID for 10 weeks.
  Interventions: Drug: Firibastat
- Group 3: ramipril 5 mg (Active Comparator): Subjects will receive 2.5 mg ramipril BID for 2 weeks and then 5 mg BID for 10 weeks.
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Ramipril — 1 or 2 capsules administered orally, twice daily
  Arms: Group 3: ramipril 5 mg
Drug: Firibastat — 1 or 2 capsules administered orally, twice daily
  Other Names: QGC001
  Arms: Group 1: firibastat 100 mg; Group 2: firibastat 500 mg

SUMMARY:
This is a multicenter, randomized, double-blind, active-controlled, dose-titrating phase 2 study to evaluate the safety and efficacy of firibastat administered orally BID (2 daily doses) versus ramipril administered orally BID over 12 weeks after acute anterior MI.

Subjects will be followed for 12 weeks (over 4 study visits). A total of 294 male and female subjects with a diagnosis of first acute anterior MI will be randomized. The subjects will need to have a primary percutaneous coronary intervention (PCI) of the index MI related artery within 24 hours after MI.

DETAILED DESCRIPTION:
At Inclusion Visit (Visit 2 [within 72 hours after acute MI]), subjects will be randomly assigned to 1 of the following 3 treatment groups in a 1:1:1 ratio:

* Group 1: Subjects will receive 50 mg firibastat BID for 2 weeks and then 100 mg BID for 10 weeks
* Group 2: Subjects will receive 250 mg firibastat BID for 2 weeks and then 500 mg BID for 10 weeks
* Group 3: Subjects will receive 2.5 mg ramipril BID for 2 weeks and then 5 mg BID for 10 weeks

Then subjects will undergo study procedures at Titration Visit (Visit 3 [Day 14]), Treatment Visit (Visit 4 Day 42]) and End-of-Treatment Visit (Visit 5 [Day 84]).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of first acute anterior MI (ST-elevation myocardial infarction) defined as chest pain >30 minutes and ST elevation ≥0.2 mV in at least 2 consecutive electrocardiogram (ECG) leads in the anterior area (DI, aVL, V1 V6).
* Primary PCI of the index-MI-related artery within 24 hours after the MI.

Exclusion Criteria:

* Body mass index >45 kg/m².
* Subject is hemodynamically unstable or has cardiogenic shock.
* Subjects with clinical signs of HF (Kilipp III and IV).
* Systolic blood pressure <100 mmHg at inclusion visit
* Early primary PCI of the index-MI-related artery performed within 3 hours after MI.
* Subjects treated with angiotensin-converting-enzyme inhibitor (ACE I), angiotensin receptor blocker (ARB) or sacubitril/valsartan prior to the index magnetic resonance imaging. Note: if treatment was for HTN, ACE I/ARB should be stopped, and, if necessary, another therapeutic class can be prescribed for HTN. If the ACE I/ARB was prescribed for congestive HF, the subject is not considered eligible; if the ACE I/ARB prescribed for another reason cannot be stopped, the subject is not eligible for study inclusion.
* Subjects scheduled for implantable cardioverter defibrillator (ICD), cardiac resynchronization therapy, or pacemaker within the next 3 months. If an ICD is indicated for ventricular arrhythmia during the course of the study, a life vest, when possible, should be prescribed and the ICD scheduled after study completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Montalescot, MD, PhD, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière - Paris
Locations (7):
- Groupe Hospitalier Pitie-Salpêtrière - Institut de Cardiologie, Paris, France
- UKSH Kiel, Kiel, Germany
- Central Hospital of Hungarian Army, Budapest, Hungary
- Krakowski Szpital Specjalistyczny im. Jana Pawła II, Krakow, Poland
- NUSCH Bratislava Dpt. of Acute Cardiology, Bratislava, Slovakia
- Hospital La Paz,, Madrid, Spain
- Freeman Hospital Newcastle upon Tyne, Newcastle, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Montalescot G, Alexander JH, Cequier-Fillat A, Solomon SD, Redheuil A, Hudec M, Silvain J, Kachenoura N, Janas A, Orban M, Josse I, Balavoine F, Besse B. Firibastat Versus Ramipril After Acute Mechanical Reperfusion of Anterior Myocardial Infarction: A Phase 2 Study. Am J Cardiovasc Drugs. 2023 Mar;23(2):207-217. doi: 10.1007/s40256-023-00567-8. Epub 2023 Feb 9. PMID 36757536
- [Derived] Khosla J, Aronow WS, Frishman WH. Firibastat: An Oral First-in-Class Brain Aminopeptidase A Inhibitor for Systemic Hypertension. Cardiol Rev. 2022 Jan-Feb 01;30(1):50-55. doi: 10.1097/CRD.0000000000000360. PMID 33027067

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 3: Ramipril 2.5 mg: Subjects will receive 5 mg ramipril BID for 2 weeks and then 5 mg BID for 10 weeks.
  Ramipril: 1 or 2 capsules administered orally, twice daily
Period: Overall Study
Arm/Group | Group 1: Firibastat 100 mg | Group 2: Firibastat 500 mg | Group 3: Ramipril 2.5 mg
Started | 98 | 99 | 98
Completed | 81 | 80 | 88
Not Completed | 17 | 19 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Firibastat 100 mg | Group 2: Firibastat 500 mg | Group 3: Ramipril 5 mg | Total
Number analyzed (Participants) | 98 | 99 | 98 | 295
Age, Categorical [Count of Participants; unit: Participants] — Population: Age analyzed on mITT population.
  Participants
    number analyzed (Participants) | 72 | 77 | 80 | 229
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 57 | 57 | 62 | 176
    >=65 years | 15 | 20 | 18 | 53
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender analyzed on mITT population
  Participants
    number analyzed (Participants) | 72 | 77 | 80 | 229
    Female | 17 | 18 | 20 | 55
    Male | 55 | 59 | 60 | 174
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hungary | 25 | 20 | 22 | 67
  Poland | 26 | 25 | 23 | 74
  United Kingdom | 1 | 2 | 2 | 5
  Slovakia | 21 | 26 | 23 | 70
  France | 13 | 14 | 13 | 40
  Germany | 4 | 3 | 4 | 11
  Spain | 8 | 9 | 11 | 28

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Ejection Fraction Assessed by Cardiac Magnetic Resonance Imaging (CMRI)
Description: Comparison of the effects of BID oral administration of 2 doses of firibastat to those of BID oral administration of ramipril on the change from Baseline in LVEF on Day 84
Time Frame: 84 days
Measure: Mean (Standard Deviation); unit: percentage of left ventricular volumes
Arm/Group | Group 1: Firibastat 100 mg | Group 2: Firibastat 500 mg | Group 3: Ramipril 5 mg
Number analyzed (Participants) | 72 | 77 | 80
percentage of left ventricular volumes | 5.6 (1.2) | 5.3 (1.1) | 5.7 (1.1)

2. Secondary Outcome: Left-ventricle End-diastolic Volume Assessed by CMRI
Description: Comparison of the effects of BID administration of firibastat and ramipril on the change from Baseline to Day 84 in left-ventricle end-diastolic volume
Time Frame: 84 days
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Group 1: Firibastat 100 mg | Group 2: Firibastat 500 mg | Group 3: Ramipril 5 mg
Number analyzed (Participants) | 72 | 77 | 80
mL | 14.2 (4.5) | 12.7 (4.3) | 9.4 (4.4)

3. Secondary Outcome: Left-ventricle End-systolic Volume Assessed by CMRI
Description: Comparison of the effects of BID administration of firibastat and ramipril on the change from Baseline to Day 84 in left-ventricle end-systolic volume
Time Frame: 84 days
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Group 1: Firibastat 100 mg | Group 2: Firibastat 500 mg | Group 3: Ramipril 5 mg
Number analyzed (Participants) | 72 | 77 | 80
mL | -0.5 (3.3) | -0.4 (3.2) | -3.1 (3.2)

4. Secondary Outcome: Major Cardiac Event (MACE): Combined Clinical Endpoint of Cardiovascular Death, MI, and Cardiac Hospitalization
Description: Comparison of the effects of BID administration of firibastat and ramipril on major cardiac event (MACE) over 84 days
Time Frame: 84 days
Measure: Number; unit: Event
Arm/Group | Group 1: Firibastat 100 mg | Group 2: Firibastat 500 mg | Group 3: Ramipril 5 mg
Number analyzed (Participants) | 98 | 98 | 98
Event | 10 | 8 | 6

5. Secondary Outcome: N-terminal Pro B-type Natriuretic Peptide (NT proBNP)
Description: Comparison of the effects of BID administration of firibastat and ramipril on the change from Baseline to Day 84 in N-terminal pro b-type natriuretic peptide (NT proBNP)
Time Frame: 84 days
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Group 1: Firibastat 100 mg | Group 2: Firibastat 500 mg | Group 3: Ramipril 5 mg
Number analyzed (Participants) | 72 | 77 | 80
pg/ml | -1618.7 (1381.7) | -1596.4 (2279.6) | -1735.6 (2326.5)

ADVERSE EVENTS:
Time Frame: Adverse events collected from the ICF signature to the end of the study.
Arm/Group | Group 1: Firibastat 100 mg | Group 2: Firibastat 500 mg | Group 3: Ramipril 5 mg
All-Cause Mortality (participants affected / at risk) | 2/98 | 1/98 | 1/98
Serious Adverse Events (participants affected / at risk) | 11/98 | 18/98 | 10/98
Other Adverse Events (participants affected / at risk) | 43/98 | 54/98 | 54/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Firibastat 100 mg (N=98) | Group 2: Firibastat 500 mg (N=98) | Group 3: Ramipril 5 mg (N=98)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Dressler's syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricule rupture (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperplasia adrenal (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal Detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain or chest discomfort (non cardiac) (General disorders) | 1 (1) | 1 (1) | 3 (3)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vascular stent trombosis (General disorders) | 1 (1) | 0 (0) | 1 (1)
COVID19 (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Staphylococcal Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Periprocedural myocadial infarction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dypsnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Firibastat 100 mg (N=98) | Group 2: Firibastat 500 mg (N=98) | Group 3: Ramipril 5 mg (N=98)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2) | 3 (4)
Coronary artery disease (Cardiac disorders) | 3 (4) | 3 (3) | 4 (4)
Dressler's syndrome (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (9) | 3 (3)
rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 4 (4) | 6 (6)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 4 (4) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Chest disconfort (General disorders) | 0 (0) | 0 (0) | 5 (5)
Chest pain (General disorders) | 2 (2) | 4 (4) | 5 (6)
Peripheral swelling (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 5 (6)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Dypsnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 2 (2) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 4 (4)
ECG QT prolonged (Investigations) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT03715998/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT03715998/SAP_001.pdf